CLINICAL TRIAL: NCT01129739
Title: Phase II Study of Umbilical Cord/Placenta-Derived Mesenchymal Stem Cells to Treat RA and RARS of MDS
Brief Title: Safety and Efficacy Study of Umbilical Cord/Placenta-Derived Mesenchymal Stem Cells to Treat Myelodysplastic Syndromes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Chengyun Zheng, Department of Hematology of the 2nd Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CZheng; No. 30670903 (Other: National Natural Science Foundation of China)
Record Dates: First submitted 2010-05-17; First posted 2010-05-25 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2010-05

CONDITIONS: Myelodysplastic Syndromes
Keywords: Bone Marrow Disease; MDS-RA; MDS-RARS; Umbilical Cord/placenta-Derived MSC; Transplant
MeSH Terms: conditions — Myelodysplastic Syndromes; Bone Marrow Diseases | interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Human umbilical cord-derived MSCs (Experimental): Human umbilical cord-derived MSCs at a dose of 1.0E+6 MSC/kg, repeated to apply in trimonthly for 2 cycle
  Interventions: Other: Human umbilical cord-derived MSCs
- cyclosporine A (CsA) (Active Comparator): CsA at a dose of 5 mg CsA/kg
  Interventions: Other: cyclosporine A (CsA)

INTERVENTIONS:
Other: Human umbilical cord-derived MSCs — 1.0E+6 MSC/kg, IV drop and repeat to apply in trimonthly for 2 cycle
  Arms: Human umbilical cord-derived MSCs
Other: cyclosporine A (CsA) — CsA 5mg/kg po for 6 months
  Arms: cyclosporine A (CsA)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of mesenchymal stem cells (MSCs) derived from human umbilical cord/placenta at a dose of 1.0E+6 MSC/kg on the subjects for refractory anemia (RA) and refractory anemia with ring sideroblast (RARS) of myelodysplastic syndromes (MDS).

DETAILED DESCRIPTION:
Myelodysplastic syndromes are bone marrow stem cell disorders resulting in disorderly and ineffective hematopoiesis. MDS is characterized by variable degrees of cytopenias (anemia, neutropenia, and thrombocytopenia ) and risk of transformation to leukemia.

To date treatment of MDS is unsatisfactory: chemotherapy has a limited role in the management of leukemic progression; autologous stem cell transplantation does not prolong relapse-free survival and stem cell transplantation is poorly tolerated in older individuals. Some MDS patients have been shown to respond to a wide variety of immunosuppressive agents ranging from corticosteroids to CsA and antithymocyte globulin (ATG). However, the overall response rate is less than 30%. In fact, few treatments appear to change the natural history of MDS.

The management of MDS patients therefore remains to be improved. Human MSCs isolated from Wharton's jelly of the umbilical cord/placenta have been shown to have immunosuppressive, stimulating hematopoiesis and tissue repairing properties. This study will evaluate the safety and effectiveness of MSC transplant in the MDS patients.

This study will last about 3 years. Participants will be randomly assigned to receive either MSC transplant (Group 1) or CsA therapy alone (Group 2). Patients will undergo MSC transplant at the start of the study (defined as Day 0). After 3 months, patients will receive the second MSC transplantation when one responds well to the treatment. After 3, 6 and 12 months from the first transplantation, patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 18~80 years old with plan to infuse MSCs.
2. Histologically documented or cytologically confirmed diagnosis of MDS with WHO classification of MDS-RA and MDS-RARS.
3. Patients must have an ECOG 0~2.
4. No moderate or sever organ dysfunction: Ejection fraction>45%; Creatinine <176 mmol/L.
5. No active severe viral or fungus infection.
6. Each patient must sign written informed consent.

Exclusion Criteria:

1. Psychiatric condition that would limit informed consent.
2. HIV positive
3. Positive Pregnancy Test
4. Patient has enrolled another clinical trial study within last 4 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
MDS clinical symptoms (mainly anemia symptoms) | 1 year
  Anemia symptoms will be mainly observed in every week after transplanting MSCs for one year.
A routine blood test | 1 year
  A routine blood test, which contains WBC, Neu, RBC, Hb and PLT, will be mainly tested in every month after transplanting MSCs for one year.
Bone borrow cytomorphologic examination | 1 year
  Bone borrow cytomorphologic examination will be tested in every 3 months after transplanting MSCs for one year.

SECONDARY OUTCOMES:
Percentage of T regulatory cell population in peripheral blood | 1 year
  Percentage of T regulatory cell population in peripheral blood will be tested in every 3 months after transplanting MSCs for one year.

CONTACTS AND LOCATIONS:
Overall Officials: cheng yun zheng, PhD, Principal Investigator — Department of Hematology of The 2nd Hospital of Shandong University
Locations (1):
- Department of Hematology of the 2nd Hospital of Shandong University, Jinan, Shandong, China